CLINICAL TRIAL: NCT04596046
Title: Comparison of the Efficiency of Systemic Therapy and Intralesional Steroid Administration in the Treatment of Idiopathic Granulomatous Mastitis
Brief Title: Could Intralesional Steroid be the Novel Treatment for Granulomatous Mastitis?
Acronym: IGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Yıldırım, Consultant General Surgeon, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95775
Record Dates: First submitted 2020-07-23; First posted 2020-10-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Granulomatous Mastitis
Keywords: Idiopathic granulomatous mastitis; intralesional steroid; systemic steroid
MeSH Terms: conditions — Granulomatous Mastitis

STUDY DESIGN:
Intervention Model Description: Prospective randomized-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S (systemic-peroral steroid) (Active Comparator): Medication of oral methylprednisolonewas administered to the patients following the adjustment based on the severity of the lesion and regarding the clinic. The prednisolone dose was 0.5 mg/kg/day in patients with painful, small (<5.0 cm) unilateral lesions whereas in multiple, bilateral lesions with the diameter of ≥5 cm or for those who had significant cutaneous ulceration, the prednisolone dose was specified as 1 mg/kg/day
  Interventions: Procedure: steroid injecting
- Group L (local-intralesional steroid) (Experimental): Triamcinolone acetonidewas administered to the patients through injecting inside the lesion. The practice was based on the dose of TCA administered in acute and chronic inflammatory skin lesions. If the lesion is single-focused and small (<5.0 cm), 20mg / mL TCA was injected and if the lesion is multifocal or large (>5.0 cm) then 40mg / mL TCA was injected into the lesion with the guidance of ultrasonography
  Interventions: Procedure: steroid injecting

INTERVENTIONS:
Procedure: steroid injecting — Group L: Triamcinolone acetonide was administered to the patients through injecting inside the lesion.Group S: Oral methylprednisolone was administered to the patients.

SUMMARY:
Idiopathic granulomatous mastitis (IGM) is a rare, benign inflammatory breast disease that mimics malignancy owing to its features of appearance.In our research, we intended to compare the efficiency of local (intralesional) steroid administration with systemic (peroral) steroid. A total of 36 patients who had been histopathologically diagnosed with IGM and whose other factors had been microbiologically excluded were included in the study. The patients were randomized into two sub-groups that would be treated with systemic and local steroids. Of the patients, 19 were administered with 0.5-1 mg/kg/day peroral systemic steroid, and 17 were administered with 40-200 mg/ml intralesional local steroid regarding the severity of the lesion. All patients were evaluated through physical examination one week after the completion of the treatment. Subsequently, the follow-up of the patients was performed thorough physical examination and ultrasonography and/or magnetic resonance imaging at the 1st, 3rd, and 6th months.

DETAILED DESCRIPTION:
The research was designed as a prospective randomized-controlled study.Prior to the study, approval was obtained from the local ethics committee of our hospital (reg.:162)The diagnosis of all patients was carried out through physical examination, imaging, and histopathology. Prior to the treatment, microbiological analysis was conducted concurrently with the biopsy.Patients who had contraindications with the use of steroids, those with active infections, as well as patients who were pregnant, and who had been diagnosed with breast cancer, were not included in the study. The patients were sub-divided into two groups as Group S (systemic-peroral steroid) and Group L (local-intralesional steroid) by using the sealed envelope randomization method. Group S: Medication of oral methylprednisolonewas administered to the patients following the adjustment based on the severity of the lesion and regarding the clinic. The prednisolone dose was 0.5 mg/kg/day in patients with painful, small (<5.0 cm) unilateral lesions whereas in multiple, bilateral lesions with the diameter of ≥5 cm or for those who had significant cutaneous ulceration, the prednisolone dose was specified as 1 mg/kg/day. Patients were informed about potential adverse effects. The medication was completed by reducing the dose. Patients in the systemic steroid group were advised to receive the medication after eating, to restrict salt and sugar consumption throughout the treatment, to quit smoking if they are using, and a proton pump inhibitor was started.Group L: Triamcinolone acetonidewas administered to the patients through injecting inside the lesion.The occurrence of systemic adverse effects in the course of the treatment was considered as the reason to discontinue the medication in all groups. Follow-up examinations of all patients at the 6th month were regarded as the endpoint of the treatment. As a consequence, it can be stated that the local (intralesional) steroid administration is also a treatment method, which is comparable to systemic steroid administration and had similar side effects. Nonetheless, it will be appropriate to promote this method by performing studies, which involve a larger population with more patients, and which is also long termed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with IGM as histopathologically

Exclusion Criteria:

* Patients who had contraindications with the use of steroids, those with active infections, as well as patients who were pregnant, and who had been diagnosed with breast cancer, were not included in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Clinical response to the treatment | 6 month
  Observational evaluation of the changes in terms of inflammation signs (hyperemia, edema, fever)
Changes in the size of the mass | 6 month
  The area of a mass captured by ultrasonography was calculated in cm^2 and the change in size was reported as a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- emine Yildirim, Gaziosmanpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Abstracts